CLINICAL TRIAL: NCT01168895
Title: Randomized, Double-blind, Cross-over Study in COPD Subjects to Investigate Safety, Tolerability, and Pharmacokinetics of Ciprofloxacin After Single Dose Inhalations of 50 mg and 75 mg Ciprofloxacin Inhalation Powder
Brief Title: Study in COPD (Chronic Obstructive Pulmonary Disease) Subjects to Investigate Safety, Tolerability, and Pharmacokinetics of Ciprofloxacin After Single Dose Inhalations of 50 mg and 75 mg Ciprofloxacin Inhalation Powder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 14972; 2010-018521-19 (EudraCT Number)
Record Dates: First submitted 2010-07-19; First posted 2010-07-23 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Infection; Pulmonary Disease, Chronic Obstructive
Keywords: 75 mg dose strength; Safety; Pharmacokinetics
MeSH Terms: conditions — Infections; Pulmonary Disease, Chronic Obstructive | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Cipro Inhale (Ciprofloxacin, BAYQ3939)
- Arm 2 (Experimental)
  Interventions: Drug: Cipro Inhale (Ciprofloxacin, BAYQ3939)

INTERVENTIONS:
Drug: Cipro Inhale (Ciprofloxacin, BAYQ3939) — 32.5 mg ciprofloxacin corresponding to 50 mg Ciprofloxacin Pulmosphere inhalation powder will be given as single dose inhalation
  Arms: Arm 1
Drug: Cipro Inhale (Ciprofloxacin, BAYQ3939) — 48.75 mg ciprofloxacin corresponding to 75 mg Ciprofloxacin Pulmosphere inhalation powder will be given as single dose inhalation
  Arms: Arm 2

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetics of ciprofloxacin after inhalation of single 52.5 and 48.75 mg doses in COPD patients. In this study the 48.75 mg dose will be administered for the first time using a new high dose strength (i.e. one capsule containing 75 mg powder = 48.75 mg ciprofloxacin) formulation. Safety investigations will focus on local tolerability in the lung and evaluate whether the patient can inhale the higher amount of powder compared to the lower dose strength. Pharmacokinetics is to see how the body absorbs, distributes, breaks down and gets rid of the study drug. Results from this study will be used to decide whether the new dose strength is suitable for larger clinical trials planned for the COPD patients population.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with COPD, 40 - 75 years of age
* All subjects must have a diagnosis of COPD and must have airway obstruction with a post-bronchodilator Forced Expiratory Volume in 1 sec (FEV1) of >/= 30% and <= 80% of predicted and a post-bronchodilator FEV1 / Forced Vital Capacity (FVC) of </= 70%
* Subjects must be current or ex-smokers with a smoking history of more than 10 pack-years
* Subjects must be able to perform technically acceptable pulmonary function tests during the study period as required in the protocol
* Subjects must be able to produce an sufficient amount of sputum during sputum induction at screening

Exclusion Criteria:

* Subjects with a significant respiratory disease other than COPD.
* Exacerbation within 8 weeks prior to screening
* Subjects with more than 1 COPD exacerbation within 12 months prior to screening
* Subjects must have an FEV1 of at least one Liter
* Subjects with a history or physician's diagnosis of asthma. If a patient has a total blood eosinophil count >/= 0.6 x 10^9/L source documentation is required to verify that the increased eosinophil count is related to a non-asthmatic condition.
* Subjects with hypersensitivity to the ciprofloxacin or to other quinolones and/or to inactive constituents of the inhalation powder
* Subjects with known hypersensitivity of the bronchial system to inhalation of nebulized drugs or saline solution
* Subjects with a history of cystic fibrosis
* Subjects with clinically evident bronchiectasis
* Subjects taking any:

  * Oral beta-adrenergic drugs or non cardioselective beta blockers,
  * Oral glucocorticoids,
  * Antihistamines or antileukotrienes prescribed for asthma,
  * Oral cromolyn sodium or oral nedocromil sodium,
  * Concomitant inhalative therapy with antibiotics and / or concomitant systemic therapy with fluoroquinolones

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Determination of ciprofloxacin pharmacokinetics derived from drug concentrations in blood, urine and sputum | Within 24 hours after treatment

SECONDARY OUTCOMES:
Adverse events collection | Within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Großhansdorf, Schleswig-Holstein, Germany